CLINICAL TRIAL: NCT05568329
Title: Appreciation for Music Processed by Hearing Aids
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, AlexanderLab, Associate Professor, Purdue University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-952
Record Dates: First submitted 2022-09-26; First posted 2022-10-05 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Sensorineural Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Hearing Aid Signal Processing (Experimental): Each subject will listen to recordings of music processed by seven different hearing aid brands set to the default "Speech in Quiet" program and the default "Music" program. Recordings (hearing aid brand x program x music sample) will be randomized from trial to trial.
  Interventions: Device: Hearing Aid Program

INTERVENTIONS:
Device: Hearing Aid Program — Each subject will listen to recordings of music processed by seven different hearing aid brands set to the default "Speech in Quiet" program and the default "Music" program. Recordings (hearing aid brand x program x music sample) will be randomized from trial to trial.
  Other Names: Hearing Aid Music Feature

SUMMARY:
Normal-hearing participants aged 18-25 with and without musical training will listen to a series of short musical samples that have been recorded through hearing aids. The music will be played at a comfortable listening level. Subjects will use the computer to rate the sound quality of the music on a 7-point Likert scale.

DETAILED DESCRIPTION:
Hearing aids are designed to treat hearing loss and restore quality of life by aiding spoken communication ability. To improve a user's listening experience for speech, hearing aids process background noise, reduce amplification for loud sounds, and use adaptive directionality for different environments, along with various other features. However, while much research and attention have been placed on developing features that improve a user's listening experience for speech, research and attention are lacking on developing features that improve a user's listening experience for music.

In addition to spoken communication, music is also influential in maintaining the quality of life. Greasley et al. (2020) report that hearing aid users, especially those who play music, often experience negative emotional consequences when they disengage from music for reasons associated with how their hearing aids amplify music. They also report that two-thirds of the hearing aid users they surveyed experienced at least some problems when listening to music. This is not a trivial issue, given that music is a significant source of entertainment - Delmonte (2018) reports that Americans aged 16 to 65+ years listen to music for more than 2 hours per day.

This study will evaluate which feature or combination of features currently being used in hearing aid music programs results in the best listening experience for music. Secondary objectives of this study will be to address the lack of information in the literature about judgments of the quality music stimuli of younger listeners, to include a wider variety of culturally inclusive music samples, and to include a comparison of preferences of musician and non-musician listeners. These objectives will be pursued by comparing the efficacy of different features used in current music programs to the default speech program and if the rankings for baseline and music features are higher or lower for musicians/non-musicians.

Participants who meet the inclusion criteria (see below) will undergo an informed consent procedure, which includes a verbal and written description of the procedures to be followed, an assurance that there are no known risks to participants, an indication of the option to withdraw from the study at any time without penalty, and the name and phone numbers of the Principal Investigator. All participants will sign the IRB-approved informed-consent form. Written consent will also be obtained for participants interested in being contacted for related studies in the future.

After informed consent, participants will complete a questionnaire about their musical experience. Participants will then have their hearing screened by an undergraduate laboratory assistant (the PI is a certified and licensed audiologist). These tests involve listening to a series of short beeps at different frequencies and intensities and pressing a button when a sound is detected. Participants who do not meet the inclusion criteria will be compensated for their time completing the questionnaire and audiologic evaluation.

During the experiments, listeners will sit in a sound-treated room and listen to brief (10-15 second) music samples presented over headphones. After each presentation, listeners will indicate their response using the computer mouse by selecting one option of a 7-point rating scale on the screen. These responses will constitute the data that will be subsequently analyzed. Sessions will last about 1 to 2 hours, including breaks taken at the participants' discretion. Data for a single experiment generally can be collected in one or two sessions, therefore, participants will be under no pressure to continue their participation over an extended period.

We will use a controlled laboratory design to investigate our questions, and participants will not have access to the sound processing outside of the laboratory. Therefore, whatever experimental manipulation we introduce immediately ceases once the participant removes the headphones.

No deception ever occurs in any of these experiments.

ELIGIBILITY:
Inclusion Criteria:

* Normal hearing (audiometric thresholds <= 20 dB HL, except one that may be 25 dB HL)
* Native English speakers

Exclusion Criteria:

-

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-21 (Actual); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-05-15 (Estimated)

PRIMARY OUTCOMES:
Sound Quality: Music Feature Activated vs. Deactivated | 60 minutes
  Within each hearing aid manufacturer, the mean sound quality with the music feature activated will be compared against the mean sound quality with the music feature deactivated.

SECONDARY OUTCOMES:
Sound Quality: Music Feature across Manufacturers | 60 minutes
  Across hearing aid manufacturers, the mean sound quality with the music feature activated will be compared.
Effects of Music Training | 60 minutes
  Mean quality ratings for subjects with more than 5 years of formal musical training will be compared against those with less than 5 years of formal musical training.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Alexander, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Data stored as a CSV file will be shared along with the audio recordings used to obtain the data. Individual participants' responses (sound quality rating) to each trial (audio recording) will be provided.
Time Frame: Upon formal acceptance of published manuscript; to be stored indefinitely.
Access Criteria: Open
URL: https://purr.purdue.edu/